CLINICAL TRIAL: NCT01314378
Title: Effects of Intensive Behavioral Training Program on Impulsivity and Inhibitory Control in Smokers
Acronym: IBTP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Massachusetts General Hospital (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH); Mind and Life Institute, Hadley, Massachusetts (Other); Harvard University (Other)
Responsible Party: Principal Investigator, Zev Schuman-Olivier, Research Fellow, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IBTP; 1R03DA030899 (NIH); 2009-1-014 (Other Grant/Funding Number: Mind and Life Institute)
Record Dates: First submitted 2011-02-24; First posted 2011-03-14 (Estimated); Last update posted 2012-05-02 (Estimated); Status verified 2012-05

CONDITIONS: Tobacco Smoking; Nicotine Dependence; Impulsivity; Addiction; Substance Dependence
Keywords: Mindfulness; Cognitive behavioral therapy; Smoking; Impulsivity; Inhibitory Control
MeSH Terms: conditions — Tobacco Smoking; Tobacco Use Disorder; Impulsive Behavior; Behavior, Addictive; Substance-Related Disorders; Smoking | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cognitive-Behavioral Therapy (Active Comparator)
  Interventions: Behavioral: Cognitive-Behavioral Therapy
- Mindfulness Training (Experimental)
  Interventions: Behavioral: Mindfulness Training

INTERVENTIONS:
Behavioral: Mindfulness Training — Eight session intensive behavioral training program for smokers
  Arms: Mindfulness Training
Behavioral: Cognitive-Behavioral Therapy — Eight session intensive behavioral intervention for smokers
  Arms: Cognitive-Behavioral Therapy

SUMMARY:
Dependence on tobacco derived nicotine is a major public health problem. Substance users who complete training in mindfulness subjectively report increased patience and improved motor control over their impulses. Yet, no studies have tested this perceived benefit with behavioral measures of impulse control. The investigators are conducting a randomized controlled clinical trial, which compares Cognitive-Behavioral Therapy and Mindfulness Training for tobacco smokers, using behavioral measures to investigate the effects of mindfulness training on impulsivity and inhibitory control.

DETAILED DESCRIPTION:
Dependence on tobacco derived nicotine is a major public health problem. Data suggest tobacco smokers are more impulsive on both self-report and behavioral measures than non-smokers. Behavioral measures of impulsivity predict outcome during smoking cessation. Successful quitters have better impulse control compared to current smokers. Impulsivity is defined behaviorally as a predisposition toward rapid, unplanned reactions to internal and external stimuli without regard for the negative consequences. Impulsivity is often measured behaviorally in two major domains, delay discounting, i.e., the choice of smaller immediate reward over a larger, delayed reward, and response inhibition, the inability to stop a response once it is initiated. A drug-free method that decreases smokers' impulsivity and enhances inhibitory control could improve sustained efficacy of smoking cessation treatment.

Treatments integrating mindfulness have been associated with decreases in impulsiveness and substance use in people with addiction. A preliminary study of reports that 100% of mindfulness-trained smokers that meditated at least 45 minutes daily were still abstinent at 6 weeks post-quit. Preliminary data suggest that mindfulness training benefits people with substance use disorders through multiple cognitive mechanisms, including decreased self-report motor impulsiveness. Yet, no widely accepted behavioral measures of impulsivity or inhibitory control have been used to measure the effect of mindfulness practice in smokers. This project aims to evaluate the relationship between mindfulness and behavioral measures of impulsivity and inhibitory control in smoking cessation and early abstinence.

Data from mindfulness-oriented treatment studies suggest at-home formal meditation practice is the most important variable in attaining positive clinical outcomes. This conclusion supports the prevailing theory that high doses of repetitive meditation practice can elicit cortical remodeling. Since addiction has been conceptualized as a disease of staged neuroplasticity, an intensive behavioral program that can induce accelerated therapeutic neuroplasticity is particularly compelling. Current methods for self-reporting dose of formal mindfulness practice may be vulnerable to response bias and poor reporting response rates. We plan to use actigraphic monitoring of formal mindfulness practice using the Actiwatch Score to behaviorally validate meditation time and rigorously test the meditation dose effect theory which hypothesizes that formal meditation practice time will predict improvement in inhibitory control, delay discounting, and smoking outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. Women and men aged 18-65, inclusive, who are competent, wish to participate and willing to provide informed consent.
2. Self report smoking >=15 cigarettes/day.
3. Expired air CO > 9ppm at the time of enrollment.

Exclusion Criteria:

1. DSM-IV diagnosis of dementia, neurodegenerative disease, or other organic mental disorder, lifetime history of psychotic disorder, bipolar disorder, severe PTSD, Dissociative Identity Disorder, OCD, anorexia nervosa, mental retardation, or autism. History of moderate or severe major depressive episode or generalized anxiety disorder within the last 6 months. Currently symptomatic ADHD with either current stimulant treatment or a history of stimulant treatment for greater than 1 year.
2. Use of prescribed psychotropic medication other than SSRI/NDRI/SNRI/buprenorphine in past 6mo, or change in such psychiatric medication dose in past six months.
3. Reported history of active substance use disorder other than nicotine or caffeine in the last six months.
4. Positive urine toxicology for illicit drugs, alcohol, opiates or benzodiazepines. (This does not include buprenorphine if participant can demonstrate 6 months of addiction treatment with negative urine screens. With the consent of the participant, participation will be discussed with the potential subject's addiction treatment provider prior to initiation of interventions.)
5. Serious unstable medical illness including, cardiovascular, hepatic, renal, respiratory, endocrine, neurological, or hematological disease such that hospitalization for treatment of that illness is likely within the next 4 months. History of life-threatening arrhythmia, CHF, syncope, or myocardial infarction within the last year. Abnormal cardiovascular event, or uncontrolled hypertension within last 2 months.
6. History of either cerebrovascular events (i.e., stroke, TIA) or head injuries with lasting neurological sequelae; history of seizure disorder or current CNS tumor.
7. Use of investigational medication in the past 30 days.
8. Third trimester pregnancy.
9. Inability to speak, read, or understand English.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2011-01; Primary Completion 2012-04 (Actual); Study Completion 2012-10 (Estimated)

PRIMARY OUTCOMES:
Expired air carbon monoxide as measure of smoking status | study week 16
  Primary Clinical Outcome Measure
Behavioral impulsivity and response inhibition as measured with Experiential Discounting Task (EDT) and Stop-Signal Task (SST). | Study week 8
  Primary Outcome Measure for Impulsivity

SECONDARY OUTCOMES:
Biochemically verified 7-day point prevalence abstinence. | Study week 16 follow-up
  Secondary Clinical Outcome Measure
Minutes of mindfulness practice will correlate with performance change in both EDT and SST. | Study week 8
  Secondary Outcome Measure for Dose Effect

CONTACTS AND LOCATIONS:
Overall Officials: Zev D Schuman-Olivier, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- MGH Center for Addiction Medicine, Boston, Massachusetts, United States

REFERENCES:
- See also: Clinical Trials at Partners Description — http://crnet.mgh.harvard.edu/trials.aspx?tId=H03846